CLINICAL TRIAL: NCT03706079
Title: A Multicentre, Double-blind, Randomized, Placebo Controlled, Parallel Group, Phase 3, Safety Extension Study to Evaluate the Safety and Tolerability of Tezepelumab in Adults and Adolescents With Severe Uncontrolled Asthma (DESTINATION)
Brief Title: Extension Study to Evaluate the Safety and Tolerability of Tezepelumab in Adults and Adolescents With Severe, Uncontrolled Asthma
Acronym: DESTINATION
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D5180C00018
Record Dates: First submitted 2018-10-11; First posted 2018-10-15 (Actual); Results first posted 2023-02-09 (Actual); Last update posted 2023-06-06 (Actual); Status verified 2023-05

CONDITIONS: Asthma
Keywords: Asthma, Uncontrolled Asthma, Severe Uncontrolled Asthma
MeSH Terms: conditions — Asthma | interventions — tezepelumab

STUDY DESIGN:
Intervention Model Description: Subjects previously randomized in one of the predecessor studies to tezepelumab will be assigned and remain on tezepelumab dosing in the Destination Study.
  Subjects randomized to placebo arm in the predecessor studies will be re-randomized in a 1:1 ratio to either tezepelumab or placebo.
  Given the randomization scheme of subjects in the predecessor studies, this will give an overall subject distribution of 3:1 (tezepelumab:placebo), assuming a similar number of subjects rollover from each arm in the predecessor studies.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double-Blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Tezepelumab (Experimental): Tezepelumab subcutaneous injection
  Interventions: Biological: Tezepelumab
- Placebo (Placebo Comparator): Placebo: Placebo subcutaneous injection
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Tezepelumab — Tezepelumab subcutaneous injection
  Arms: Tezepelumab
Other: Placebo — Placebo subcutaneous injection
  Arms: Placebo

SUMMARY:
Subjects who completed either D5180C00007 or D5180C00009 will be offered the opportunity to consent for the Multicentre, Double-blind, Randomized, Placebo Controlled, Parallel Group, Phase 3, Safety Extension Study to Evaluate the Safety and Tolerability of Tezepelumab in Adults and Adolescents with Severe Uncontrolled Asthma. The study consists of a treatment phase, followed by a follow-up phase where subjects will not receive IP. The length of the follow up phase is determined by which study the subject had previously completed.

DETAILED DESCRIPTION:
Subjects who have not met investigational product discontinuation criteria and have attended the EOT visit in either study D5180C00007 or D5180C00009 will be offered the opportunity to consent for the Multicentre, Double-blind, Randomized, Parallel Group, Placebo Controlled, Phase 3, Safety Extension Study to Evaluate the Safety and Tolerability of Tezepelumab versus placebo in Adults and Adolescents (12 years of age and older) with a history of asthma exacerbations and inadequately controlled severe asthma receiving medium or high dose inhaled corticosteroid (ICS) plus at least one additional asthma controller medication with or without oral corticosteroids

Following treatment, subjects will enter a follow-up phase, determined by the predecessor study they had previously completed. Subjects will not receive IP during the follow-up phase. For subjects who entered the study from study D5180C00007 and did not meet IP Discontinuation criteria, the follow-up phase will extend from week 104 to Week 140. Subjects who entered the study from study D5180C00009 will have their follow-up phase extend to week 116.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated written informed consent
* Negative urine test for female subjects of childbearing potential prior to administration of IP at visit 1
* Females of childbearing potential who are sexually active with a nonsterilized male partner must use a highly effective method of contraception from screening, and must agree to continue using such precautions for 16 weeks after the final dose of IP.
* Female or male subjects who have not met investigational product discontinuation criteria and have attended the EOT visit in either study D5180C00007 (NAVIGATOR) or D5180C00009 (SOURCE)

To enter the extended follow-up phase of the study, the following inclusion criteria also apply:

* Provision of signed and dated Addendum for Extended Follow-up to informed consent, as well as assent by adolescent subjects where applicable, prior to any mandatory study specific procedures, sampling and analyses before Extended Follow Up.
* Must have entered DESTINATION from D5180C00007 study and have completed IP dosing to Week 100, have not met IP Discontinuation criteria and have attended the EOT Visit.

Exclusion Criteria:

* Any clinically important pulmonary disease other than asthma
* Any disorder, including, but not limited to cardiovascular, gastrointestinal, hepatic, renal, neurological, musculoskeletal, infectious, endocrine, metabolic, hematological, psychiatric, or major physical impairment that is not stable
* History of chronic alcohol or drug abuse within 12 months prior to visit 1
* Current malignancy or malignancy that developed during a predecessor study
* Major surgery or planned surgical procedures requiring general anesthesia or inpatient status for > 1 day during the conduct of the study
* Treatment with systemic immunosuppressive/immunomodulating drugs except for OCS used in the treatment of asthma/asthma exacerbations within the last 12 weeks prior to randomization
* Concurrent enrolment in another clinical study involving an IP
* Any clinically meaningful abnormal finding in physical examination, vital signs, ECG,haematology, clinical chemistry, or urinalysis during the predecessor study
* Pregnant, breastfeeding, or lactating

To enter the extended follow-up phase of the study (which extends from week 104 to week 140), the following exclusion criteria also apply:

* Discontinuation of IP during the treatment period of DESTINATION.
* Entered DESTINATION from D5180C00009 (SOURCE) study.

Ages: 13 Years to 81 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 951 (Actual)
Dates: Start 2019-01-07 (Actual); Primary Completion 2021-10-26 (Actual); Study Completion 2022-05-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Menzies-Gow, MD, Principal Investigator — Royal Brompton Hospital, United Kingdom
Locations (147):
- United States (48):
  - Research Site, Dothan, Alabama
  - Research Site, Gilbert, Arizona
  - Research Site, Bakersfield, California
  - Research Site, Huntington Beach, California
  - Research Site, Long Beach, California
  - Research Site, Los Angeles, California
  - Research Site, Newport Beach, California
  - Research Site, Northridge, California
  - Research Site, Palm Desert, California
  - Research Site, Rolling Hills Estates, California
  - Research Site, Walnut Creek, California
  - Research Site, Westminster, California
  - Research Site, New Haven, Connecticut
  - Research Site, Kissimmee, Florida
  - Research Site, Port Charlotte, Florida
  - Research Site, Sarasota, Florida
  - Research Site, Tampa, Florida
  - Research Site, Winter Park, Florida
  - Research Site, Boise, Idaho
  - Research Site, Zachary, Louisiana
  - Research Site, White Marsh, Maryland
  - Research Site, Boston, Massachusetts
  - Research Site, Ann Arbor, Michigan
  - Research Site, St Louis, Missouri
  - Research Site, Lincoln, Nebraska
  - Research Site, Las Vegas, Nevada
  - Research Site, Northfield, New Jersey
  - Research Site, Brooklyn, New York
  - Research Site, The Bronx, New York
  - Research Site, Charlotte, North Carolina
  - Research Site, Durham, North Carolina
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Cincinnati, Ohio
  - Research Site, Edmond, Oklahoma
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Medford, Oregon
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Anderson, South Carolina
  - Research Site, Columbia, South Carolina
  - Research Site, Greenville, South Carolina
  - Research Site, Amarillo, Texas
  - Research Site, Boerne, Texas
  - Research Site, McKinney, Texas
  - Research Site, Plano, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Manassas, Virginia
  - Research Site, Cudahy, Wisconsin
  - Research Site, Madison, Wisconsin
- Argentina (9):
  - Research Site, Buenos Aires
  - Research Site, CABA
  - Research Site, Ciudad de Buenos Aires
  - Research Site, Córdoba
  - Research Site, Mendoza
  - Research Site, Nueve de Julio
  - Research Site, Quilmes
  - Research Site, San Fernando
  - Research Site, San Miguel de Tucumán
- Australia (6):
  - Research Site, Kent Town
  - Research Site, Melbourne
  - Research Site, New Lambton
  - Research Site, Spearwood
  - Research Site, Westmead
  - Research Site, Woolloongabba
- Research Site, Vienna, Austria
- Brazil (9):
  - Research Site, Blumenau
  - Research Site, Botucatu
  - Research Site, Curitiba
  - Research Site, Porto Alegre
  - Research Site, Recife
  - Research Site, Salvador
  - Research Site, Santo André
  - Research Site, São Bernardo do Campo
  - Research Site, Sorocaba
- Canada (10):
  - Research Site, Calgary, Alberta
  - Research Site, Sherwood Park, Alberta
  - Research Site, Ajax, Ontario
  - Research Site, Mississauga, Ontario
  - Research Site, Ottawa, Ontario
  - Research Site, Windsor, Ontario
  - Research Site, Montreal, Quebec
  - Research Site, Québec, Quebec
  - Research Site, Saint-Charles-Borromée, Quebec
  - Research Site, Trois-Rivières, Quebec
- France (9):
  - Research Site, Brest
  - Research Site, Le Kremlin-Bicêtre
  - Research Site, Lyon
  - Research Site, Marseille
  - Research Site, Montpellier
  - Research Site, Nantes
  - Research Site, Paris
  - Research Site, Pessac
  - Research Site, Strasbourg
- Germany (11):
  - Research Site, Bamberg
  - Research Site, Berlin
  - Research Site, Frankfurt
  - Research Site, Frankfurt am Main
  - Research Site, Hamburg
  - Research Site, Hanover
  - Research Site, Koblenz
  - Research Site, Landsberg
  - Research Site, Leipzig
  - Research Site, Lübeck
  - Research Site, Mainz
- Israel (5):
  - Research Site, Ashkelon
  - Research Site, Haifa
  - Research Site, Jerusalem
  - Research Site, Kfar Saba
  - Research Site, Rehovot
- Poland (3):
  - Research Site, Krakow
  - Research Site, Lodz
  - Research Site, Wroclaw
- Russia (3):
  - Research Site, Izhevsk
  - Research Site, Moscow
  - Research Site, Saint Petersburg
- Research Site, Jeddah, Saudi Arabia
- South Africa (9):
  - Research Site, Bellville
  - Research Site, Cape Town
  - Research Site, Durban
  - Research Site, eMkhomazi
  - Research Site, Johannesburg
  - Research Site, Lenasia Ext8
  - Research Site, Meadowdale, Germiston
  - Research Site, Middelburg
  - Research Site, Parow
- South Korea (8):
  - Research Site, Bucheon-si
  - Research Site, Cheongju-si
  - Research Site, Daegu
  - Research Site, Jeju-do
  - Research Site, Jeonju
  - Research Site, Seongnam-si
  - Research Site, Seoul
  - Research Site, Suwon
- Taiwan (3):
  - Research Site, Kaohsiung City
  - Research Site, Taichung
  - Research Site, Taipei
- Turkey (Türkiye) (3):
  - Research Site, Ankara
  - Research Site, Bursa
  - Research Site, Istanbul
- Ukraine (6):
  - Research Site, Dnipro
  - Research Site, Ivano-Frankivsk
  - Research Site, Kharkiv Region
  - Research Site, Kherson
  - Research Site, Lutsk
  - Research Site, Vinnytsia
- Vietnam (3):
  - Research Site, Hanoi
  - Research Site, Hà Nội
  - Research Site, Ho Chi Minh City

REFERENCES:
- [Derived] Wechsler ME, Brusselle G, Virchow JC, Bourdin A, Kostikas K, Llanos JP, Roseti SL, Ambrose CS, Hunter G, Jackson DJ, Castro M, Lugogo N, Pavord ID, Martin N, Brightling CE. Clinical response and on-treatment clinical remission with tezepelumab in a broad population of patients with severe, uncontrolled asthma: results over 2 years from the NAVIGATOR and DESTINATION studies. Eur Respir J. 2024 Dec 5;64(6):2400316. doi: 10.1183/13993003.00316-2024. Print 2024 Dec. PMID 39326921
- [Derived] Brightling CE, Caminati M, Llanos JP, Caveney S, Kotalik A, Griffiths JM, Lundahl A, Israel E, Pavord ID, Wechsler ME, Porsbjerg C, Corren J, Golabek M, Martin N, Ponnarambil S. Biomarkers and clinical outcomes after tezepelumab cessation: Extended follow-up from the 2-year DESTINATION study. Ann Allergy Asthma Immunol. 2024 Sep;133(3):310-317.e4. doi: 10.1016/j.anai.2024.04.031. Epub 2024 Apr 30. PMID 38697286
- [Derived] Menzies-Gow A, Wechsler ME, Brightling CE, Korn S, Corren J, Israel E, Chupp G, Bednarczyk A, Ponnarambil S, Caveney S, Almqvist G, Golabek M, Simonsson L, Lawson K, Bowen K, Colice G; DESTINATION study investigators. Long-term safety and efficacy of tezepelumab in people with severe, uncontrolled asthma (DESTINATION): a randomised, placebo-controlled extension study. Lancet Respir Med. 2023 May;11(5):425-438. doi: 10.1016/S2213-2600(22)00492-1. Epub 2023 Jan 23. PMID 36702146
- [Derived] Menzies-Gow A, Ponnarambil S, Downie J, Bowen K, Hellqvist A, Colice G. DESTINATION: a phase 3, multicentre, randomized, double-blind, placebo-controlled, parallel-group trial to evaluate the long-term safety and tolerability of tezepelumab in adults and adolescents with severe, uncontrolled asthma. Respir Res. 2020 Oct 21;21(1):279. doi: 10.1186/s12931-020-01541-7. PMID 33087119
- See also: Statistical Analysis Plan (SAP) — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5180C00018&attachmentIdentifier=8a2b972e-4a6e-43c5-af7a-ae92fb0c49f3&fileName=d5180c00018-sap-ed-3-redact.pdf&versionIdentifier=
- See also: Protocol — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5180C00018&attachmentIdentifier=50cb4a27-8cdd-456e-8557-fdeccbd69d40&fileName=d5180c00018-csp-v6-redact.pdf&versionIdentifier=
- See also: CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5180C00018&attachmentIdentifier=d7be4478-ea53-4972-9b54-6771c586611a&fileName=d5180c00018-study-synopsis-redact.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants who completed treatment and attended end of treatment visit in predecessor studies NAVIGATOR (NCT03347279) or SOURCE (NCT03406078) were eligible for this long-term extension study. In the predecessor studies, a total of 1059 and 150 subjects were randomised and dosed in NAVIGATOR and SOURCE respectively. In DESTINATION, a total of 951 subjects (827 from NAVIGATOR and 124 from SOURCE) were randomised at 182 centres in 18 countries to receive treatment with tezepelumab or placebo.
Pre-assignment Details: Of the 1209 patients randomized and dosed in predecessor studies, 951 were randomised in DESTINATION and 950 received treatment. The patients receiving tezepelumab in the predecessors continued to receive tezepelumab, while patients receiving placebo in the predecessors were re-randomized 1:1 to either receive tezepelumab in DESTINATION or to continue placebo, resulting in a 3:1 randomization ratio in DESTINATION.
Groups:
- NAVIGATOR Rand Teze: All subjects randomised to tezepelumab in the NAVIGATOR predecessor and treated with at least one dose in the predecessor, regardless of whether they participated in the DESTINATION study.
- NAVIGATOR Rand Pbo: All subjects randomised to placebo in the NAVIGATOR predecessor and treated with at least one dose in the predecessor, regardless of whether they participated in the DESTINATION study. For subjects switching to tezepelumab in DESTINATION, data collected during the placebo (predecessor) period are contained in this column, while data collected after the first dose of tezepelumab in DESTINATION are presented in the NAVIGATOR Pbo to Teze arm.
- NAVIGATOR Pbo to Teze: All subjects randomised to placebo in the NAVIGATOR predecessor and re-randomised to tezepelumab in DESTINATION. Only data collected after the first dose of tezepelumab in DESTINATION are presented in this column.
- SOURCE Rand Teze: All subjects randomised to tezepelumab in the SOURCE predecessor and treated with at least one dose in the predecessor, regardless of whether they participated in the DESTINATION study.
- SOURCE Rand Pbo: All subjects randomised to placebo in the SOURCE predecessor and treated with at least one dose in the predecessor, regardless of whether they participated in the DESTINATION study. For subjects switching to tezepelumab in DESTINATION, data collected during the placebo (predecessor) period are contained in this column, while data collected after the first dose of tezepelumab in DESTINATION are presented in the SOURCE Pbo to Teze arm.
- SOURCE Pbo to Teze: All subjects randomised to placebo in the SOURCE predecessor and re-randomised to tezepelumab in DESTINATION. Only data collected after the first dose of tezepelumab in DESTINATION are presented in this column.
Period: Predecessor Study
Arm/Group | NAVIGATOR Rand Teze | NAVIGATOR Rand Pbo | NAVIGATOR Pbo to Teze | SOURCE Rand Teze | SOURCE Rand Pbo | SOURCE Pbo to Teze
Started | 529 | 532 | 0 (Not Applicable for predecessor period) | 74 | 76 | 0 (Not Applicable for predecessor period)
Received Treatment | 528 | 531 | 0 (Not Applicable for predecessor period) | 74 | 76 | 0 (Not Applicable for predecessor period)
Completed | 513 | 509 | 0 (Not Applicable for predecessor period) | 68 | 73 | 0 (Not Applicable for predecessor period)
Not Completed | 16 | 23 | 0 | 6 | 3 | 0
Not completed — Death | 0 | 2 | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 5 | 2 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 8 | 15 | 0 | 5 | 2 | 0
Not completed — Did not receive treatment / Non-compliance with protocol / did not complete safety follow-up visits | 3 | 4 | 0 | 0 | 0 | 0
Period: Long Term Extension (DESTINATION)
Arm/Group | NAVIGATOR Rand Teze | NAVIGATOR Rand Pbo | NAVIGATOR Pbo to Teze | SOURCE Rand Teze | SOURCE Rand Pbo | SOURCE Pbo to Teze
Started | 415 | 206 | 206 | 60 | 32 | 32
Received Treatment | 415 | 206 | 205 | 60 | 32 | 32
Completed | 400 | 200 | 198 | 58 | 28 | 31
Not Completed | 15 | 6 | 8 | 2 | 4 | 1
Not completed — Due to COVID-19 pandemic | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Did not complete safety follow-up visits | 1 | 0 | 2 | 0 | 0 | 0
Not completed — Pregnancy | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 3 | 3 | 1 | 3 | 0
Not completed — Lost to Follow-up | 2 | 1 | 1 | 0 | 1 | 0
Not completed — Death | 8 | 2 | 2 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- NAVIGATOR Rand Pbo: All subjects randomised to placebo in the NAVIGATOR predecessor and treated with at least one dose in the predecessor, regardless of whether they participated in the DESTINATION study and regardless of their treatment assignment in DESTINATION.
- SOURCE Rand Pbo: All subjects randomised to placebo in the SOURCE predecessor and treated with at least one dose in the predecessor, regardless of whether they participated in the DESTINATION study and regardless of their treatment assignment in DESTINATION.
- Total: Total of all reporting groups
Arm/Group | NAVIGATOR Rand Teze | NAVIGATOR Rand Pbo | SOURCE Rand Teze | SOURCE Rand Pbo | Total
Number analyzed (Participants) | 528 | 531 | 74 | 76 | 1209
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 41 | 41 | 0 | 0 | 82
  Between 18 and 65 years | 391 | 416 | 58 | 62 | 927
  >=65 years | 96 | 74 | 16 | 14 | 200
Age, Continuous [Mean (Standard Deviation); unit: Years] | 49.9 (16.3) | 49.0 (15.9) | 53.5 (12.1) | 53.4 (11.9) | 49.9 (15.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 335 | 337 | 49 | 45 | 766
  Male | 193 | 194 | 25 | 31 | 443
Race/Ethnicity, Customized [Number; unit: Participants]
  Hispanic or Latino | 83 | 81 | 10 | 14 | 188
  Not Hispanic or Latino | 445 | 450 | 64 | 62 | 1021
Race/Ethnicity, Customized [Number; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 0 | 1
  Asian | 146 | 149 | 11 | 11 | 317
  Black of African American | 30 | 31 | 1 | 0 | 62
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 0 | 1
  Other | 19 | 23 | 0 | 1 | 43
  White | 332 | 327 | 62 | 64 | 785

OUTCOME MEASURES:

1. Secondary Outcome: Annualized Asthma Exacerbation Rate (AAER)
Description: The annualized exacerbation rate is based on exacerbations reported by the investigator in the eCRF. The analysis is based on the primary population (Full Analysis Set)
Time Frame: Baseline (Week 0 in predecessor study) to Week 104. For subjects switching treatments from placebo in the predecessor to tezepelumab in DESTINATION, all data collected after first dose of tezepelumab are excluded.
Measure: Least Squares Mean (95% Confidence Interval); unit: events per year
Groups:
- NAVIGATOR Rand Pbo: All subjects randomised to placebo in the NAVIGATOR predecessor and treated with at least one dose in the predecessor, regardless of whether they participated in the DESTINATION study. For subjects switching treatments from placebo in the predecessor to tezepelumab in DESTINATION, all data collected after first dose of tezepelumab are excluded.
- SOURCE Rand Pbo: All subjects randomised to placebo in the SOURCE predecessor and treated with at least one dose in the predecessor, regardless of whether they participated in the DESTINATION study. For subjects switching treatments from placebo in the predecessor to tezepelumab in DESTINATION, all data collected after first dose of tezepelumab are excluded.
Arm/Group | NAVIGATOR Rand Teze | NAVIGATOR Rand Pbo | SOURCE Rand Teze | SOURCE Rand Pbo
Number analyzed (Participants) | 528 | 531 | 74 | 76
events per year | 0.82 [0.71 to 0.95] | 1.93 [1.70 to 2.20] | 1.07 [0.76 to 1.51] | 1.76 [1.27 to 2.45]
Statistical Analysis 1: Comparison: NAVIGATOR Rand Teze vs NAVIGATOR Rand Pbo; Test type: Superiority; Rate Ratio = 0.42, 95% CI 2-sided [0.35 to 0.51]
Statistical Analysis 2: Comparison: SOURCE Rand Teze vs SOURCE Rand Pbo; Test type: Superiority; Rate Ratio = 0.61, 95% CI 2-sided [0.38 to 0.96]

2. Primary Outcome: Exposure Adjusted Incidence Rates of AEs/SAEs
Description: Includes adverse events with an onset date between the date of first dose of IP in the predecessor and minimum (date of last dose of IP + 33 days, date of death, date of study withdrawal, day prior to start of another biologic). The analysis is based on the Safety Analysis Set. Exposure adjusted rates are defined as number of subjects with AEs divided by total time at risk across all subjects, multiplied by 100
Time Frame: as for outcome 1
Measure: Number; unit: Patients with AEs per 100 person-years
Arm/Group | NAVIGATOR Rand Teze | NAVIGATOR Rand Pbo | SOURCE Rand Teze | SOURCE Rand Pbo
Number analyzed (Participants) | 528 | 531 | 74 | 76
Patients with AEs per 100 person-years
  Any AE incidence rate | 49.62 | 62.66 | 47.15 | 69.97
  Any AE with outcome=death incidence rate | 0.76 | 0.14 | 1.55 | 0.00
  Any SAE incidence rate | 7.85 | 12.45 | 13.14 | 17.99
  Any AE leading to discontinuation of IP incidence rate | 1.64 | 3.00 | 1.55 | 2.00

3. Primary Outcome: Total Time at Risk
Description: Includes time between the date of first dose of IP in the predecessor and minimum (date of last dose of IP + 33 days, date of death, date of study withdrawal, day prior to start of another biologic). The analysis is based on the Safety Analysis Set.
Time Frame: as for outcome 1
Measure: Number; unit: Year
Arm/Group | NAVIGATOR Rand Teze | NAVIGATOR Rand Pbo | SOURCE Rand Teze | SOURCE Rand Pbo
Number analyzed (Participants) | 528 | 531 | 74 | 76
Year | 917.0 | 699.0 | 129.4 | 100.0

ADVERSE EVENTS:
Time Frame: Baseline (Week 0 in predecessor study) to long-term extension completion (either weeks 104 or 116). Includes AEs with onset date between the date of first dose of IP and and the long-term extension completion or withdrawal date (on-study period)
Description: The subjects switching treatments from placebo in the predecessor to tezepelumab in DESTINATION are included in both Rand Pbo and Pbo to Teze arms. Their data collected during the placebo (predecessor) period are contained within the Rand Pbo arm, while data collected after the first dose of tezepelumab in DESTINATION are presented in the Pbo to Teze arm. Note the primary objective in the Outcome Measures section presents on-treatment safety as opposed to on-study safety.
Arm/Group | NAVIGATOR Rand Teze | NAVIGATOR Rand Pbo | NAVIGATOR Pbo to Teze | SOURCE Rand Teze | SOURCE Rand Pbo | SOURCE Pbo to Teze
All-Cause Mortality (participants affected / at risk) | 8/528 | 5/531 | 1/206 | 2/74 | 0/76 | 0/32
Serious Adverse Events (participants affected / at risk) | 82/528 | 94/531 | 17/206 | 18/74 | 19/76 | 4/32
Other Adverse Events (participants affected / at risk) | 390/528 | 384/531 | 98/206 | 53/74 | 58/76 | 23/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NAVIGATOR Rand Teze (N=528) | NAVIGATOR Rand Pbo (N=531) | NAVIGATOR Pbo to Teze (N=206) | SOURCE Rand Teze (N=74) | SOURCE Rand Pbo (N=76) | SOURCE Pbo to Teze (N=32)
Cardiac failure congestive (Cardiac disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Periprocedural myocardial infarction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coronary artery occlusion (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ulna fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ligament rupture (Injury, poisoning and procedural complications) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle necrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocarditis (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gout (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Amyotrophy (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bone cyst (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Exostosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Invasive breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Polyarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Prinzmetal angina (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Encephalocele (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Immune thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertrophic cardiomyopathy (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertigo positional (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 1 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anal fistula (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Uveitis (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diverticular perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute left ventricular failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastric polyps (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ileus paralytic (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 2 (3) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oesophageal achalasia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis necrotising (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Death (General disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Impaired healing (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aortic valve stenosis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis chronic (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Drug-induced liver injury (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breast abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bacterial pyelonephritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Covid-19 (Infections and infestations) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Covid-19 pneumonia (Infections and infestations) | 3 (3) | 2 (2) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
H1n1 influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intervertebral discitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lower respiratory tract infection bacterial (Infections and infestations) | 0 (0) | 2 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Meningitis bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 3 (3) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia haemophilus (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Osteomyelitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia streptococcal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Periorbital cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (2) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Pneumonia klebsiella (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ovarian germ cell teratoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Benign neoplasm of thyroid gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colon cancer stage iv (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neurilemmoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Squamous cell carcinoma of the oral cavity (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thymoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Glomerulonephritis membranous (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal colic (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cubital tunnel syndrome (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhagic stroke (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 14 (18) | 41 (79) | 5 (6) | 3 (5) | 8 (11) | 0 (0)
Idiopathic generalised epilepsy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intracranial aneurysm (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lumbar radiculopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Migraine (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myelopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ruptured cerebral aneurysm (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Disruptive mood dysregulation disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Obstruction gastric (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atypical pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis infective (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster oticus (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis salmonella (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Septic shock (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Incisional hernia (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bipolar disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Uterine prolapse (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 16 (20) | 43 (91) | 5 (6) | 5 (7) | 8 (12) | 0 (0)
Bronchial secretion retention (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eosinophilic pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary sarcoidosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperparathyroidism primary (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cyanosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis ischaemic (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis chronic (Hepatobiliary disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anal abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia aspiration (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia staphylococcal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NAVIGATOR Rand Teze (N=528) | NAVIGATOR Rand Pbo (N=531) | NAVIGATOR Pbo to Teze (N=206) | SOURCE Rand Teze (N=74) | SOURCE Rand Pbo (N=76) | SOURCE Pbo to Teze (N=32)
Sinusitis (Infections and infestations) | 30 (34) | 43 (64) | 5 (5) | 2 (2) | 5 (6) | 1 (1)
Traumatic haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Rhinitis (Infections and infestations) | 18 (24) | 21 (42) | 6 (26) | 4 (4) | 2 (2) | 0 (0)
Sinusitis bacterial (Infections and infestations) | 2 (2) | 1 (1) | 1 (1) | 5 (5) | 1 (1) | 0 (0)
Upper respiratory tract infection bacterial (Infections and infestations) | 8 (10) | 2 (6) | 1 (1) | 3 (3) | 1 (1) | 0 (0)
Vaginal infection (Infections and infestations) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperlipidaemia (Metabolism and nutrition disorders) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 16 (16) | 8 (9) | 3 (3) | 1 (1) | 2 (2) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 36 (49) | 25 (30) | 5 (5) | 3 (4) | 2 (2) | 0 (0)
Vertebral foraminal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyposmia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Spinal cord disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 11 (13) | 8 (9) | 5 (5) | 0 (0) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 15 (15) | 8 (9) | 2 (3) | 2 (2) | 2 (2) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 9 (9) | 8 (9) | 2 (2) | 3 (3) | 2 (3) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Acute sinusitis (Infections and infestations) | 16 (23) | 16 (26) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Bronchitis bacterial (Infections and infestations) | 30 (34) | 19 (24) | 3 (3) | 8 (20) | 7 (10) | 3 (5)
Bronchitis viral (Infections and infestations) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 2 (3) | 2 (2)
Oral candidiasis (Infections and infestations) | 12 (16) | 15 (17) | 2 (2) | 5 (6) | 6 (11) | 2 (2)
Pharyngitis (Infections and infestations) | 26 (35) | 23 (28) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Pneumonia haemophilus (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Suspected covid-19 (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Tinea versicolour (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 72 (131) | 91 (151) | 6 (7) | 12 (13) | 9 (9) | 0 (0)
Urinary tract infection (Infections and infestations) | 29 (50) | 29 (33) | 9 (10) | 1 (1) | 1 (2) | 2 (2)
Viral rhinitis (Infections and infestations) | 7 (7) | 4 (4) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 24 (31) | 17 (23) | 5 (5) | 2 (5) | 3 (3) | 2 (2)
Vulval abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 14 (20) | 9 (10) | 2 (2) | 3 (4) | 1 (1) | 0 (0)
Facial bones fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 9 (9) | 12 (12) | 4 (4) | 3 (3) | 4 (4) | 2 (2)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 12 (14) | 9 (9) | 5 (5) | 1 (1) | 1 (1) | 1 (1)
Glucose tolerance impaired (Metabolism and nutrition disorders) | 3 (3) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 27 (46) | 21 (23) | 3 (3) | 2 (2) | 3 (4) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 12 (15) | 11 (13) | 1 (1) | 5 (7) | 1 (2) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 18 (21) | 11 (12) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 5 (6) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anosmia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cerebral arteriosclerosis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cerebrovascular disorder (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 58 (157) | 54 (101) | 13 (18) | 9 (16) | 10 (12) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 14 (17) | 25 (27) | 2 (3) | 6 (7) | 9 (16) | 0 (0)
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (6) | 0 (0) | 1 (1) | 5 (7) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 30 (39) | 22 (31) | 3 (5) | 0 (0) | 0 (0) | 1 (1)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 6 (6) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 4 (4) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Photodermatosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (4) | 9 (12) | 1 (2) | 3 (3) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 7 (7) | 7 (7) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Rash macular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 30 (39) | 26 (40) | 4 (4) | 5 (7) | 7 (7) | 4 (4)
Cataract (Eye disorders) | 7 (8) | 2 (3) | 0 (0) | 2 (2) | 3 (3) | 1 (1)
Retinal tear (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dental caries (Gastrointestinal disorders) | 3 (3) | 6 (6) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 7 (13) | 4 (4) | 1 (2) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 16 (19) | 9 (10) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Impaired healing (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Influenza like illness (General disorders) | 26 (28) | 25 (29) | 5 (6) | 0 (0) | 6 (6) | 0 (0)
Pyrexia (General disorders) | 12 (12) | 9 (11) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 29 (44) | 39 (51) | 2 (2) | 9 (10) | 3 (3) | 0 (0)
Covid-19 (Infections and infestations) | 7 (8) | 8 (8) | 10 (10) | 5 (5) | 1 (1) | 4 (4)
Chronic sinusitis (Infections and infestations) | 9 (13) | 6 (8) | 1 (1) | 3 (4) | 4 (4) | 0 (0)
Cystitis (Infections and infestations) | 8 (9) | 9 (11) | 1 (1) | 0 (0) | 1 (2) | 1 (2)
Gastroenteritis (Infections and infestations) | 25 (26) | 16 (17) | 5 (5) | 2 (2) | 1 (1) | 0 (0)
Lower respiratory tract infection bacterial (Infections and infestations) | 9 (11) | 8 (10) | 3 (4) | 1 (1) | 1 (1) | 1 (2)
Nasopharyngitis (Infections and infestations) | 130 (220) | 124 (222) | 21 (26) | 18 (27) | 22 (38) | 7 (12)
Otitis media (Infections and infestations) | 10 (12) | 4 (4) | 2 (2) | 0 (0) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-04-12): https://cdn.clinicaltrials.gov/large-docs/79/NCT03706079/Prot_000.pdf
  • Statistical Analysis Plan (2021-11-03): https://cdn.clinicaltrials.gov/large-docs/79/NCT03706079/SAP_001.pdf